CLINICAL TRIAL: NCT03422393
Title: A Phase 1 Clinical Trial to Evaluate Venetoclax With High-dose Ibrutinib for the Treatment of Patients With Chronic Lymphocytic Leukemia With Progressive Disease on Single Agent Ibrutinib.
Brief Title: Venetoclax With High-dose Ibrutinib for CLL Progressing on Single Agent Ibrutinib
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Choi (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Michael Choi, Clinical investigator, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 171613
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: venetoclax; ibrutinib; high-dose ibrutinib; chronic lymphocytic leukemia; progressive disease; Small Lymphocytic Lymphoma; cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Disease Progression; Neoplasms | interventions — venetoclax; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- venetoclax with high-dose ibrutinib (Experimental): venetoclax with high-dose ibrutinib for the treatment of patients with chronic lymphocytic leukemia with progressive disease on single agent ibrutinib.
  Interventions: Drug: Venetoclax; Drug: Ibrutinib

INTERVENTIONS:
Drug: Venetoclax — On cycle 1, day 1, patients will initiate venetoclax. The dose of venetoclax will ramp-up from 20 mg PO daily to 400 mg PO daily over a 5 week period.
  Other Names: Venclexta
Drug: Ibrutinib — During the screening period, patients will continue on ibrutinib at their previous tolerated dose, unless required to stop (e.g.: by a preceding clinical trial).
  On cycle 1, day 1, the dose of ibrutinib will be assigned based on the dose cohort. Patients in cohort 1 will receive ibrutinib 420 mg PO daily. Patients in cohort 2 will receive ibrutinib 560 mg PO daily. Cohort 3 will be 840 mg PO daily.
  Other Names: Imbruvica

SUMMARY:
The purpose of the study is to investigate whether the combination of venetoclax and ibrutinib (administered up to 840 mg per day) might be useful for the treatment of CLL or SLL that is not responding or no longer responding to treatment with ibrutinib alone. The study will evaluate whether this regimen can reduce the amount of cancerous cells in your body. If you agree, you will receive ibrutinib at a dose of up to 840 mg a day by mouth, as well as venetoclax. Although both of these agents are approved by the FDA for the treatment of CLL or SLL, the combination and the dosing schedule of ibrutinib are considered experimental.

DETAILED DESCRIPTION:
This is phase 1 study for patients with CLL or small lymphocytic lymphoma (SLL) experiencing disease progression on single ibrutinib. This study will evaluate the optimal ibrutinib dose (including doses higher than 420 mg) when combined with venetoclax

During the screening period, patients will continue on ibrutinib at their previous tolerated dose, unless required to stop (e.g.: by a preceding clinical trial).

On cycle 1, day 1, the dose of ibrutinib will be assigned based on the dose cohort. Patients in cohort 1 will receive ibrutinib 420 mg PO daily. Patients in cohort 2 will receive ibrutinib 560 mg PO daily. Cohort 3 will be 840 mg PO daily.

On cycle 1, day 1, patients will initiate venetoclax. The dose of venetoclax will ramp-up from 20 mg PO daily to 400 mg PO daily over a 5 week period.

The primary safety endpoint is determination of DLTs during the first 35 days (completion of dose ramp up). The primary efficacy endpoint of overall response rate will be assessed on approximately Cycle 7, Day 1.

Rationale: The optimal management of patients that progress on ibrutinib, including those with acquired Btk or PLCg2 mutations, is not determined. In other cancers, continued treatment with small molecule inhibitors beyond disease progression provides significant benefit, with additional agents or adjustments to ablate the resistant subclone. Venetoclax is approved for the treatment of patients with CLL, and is well-tolerated and effective in high-risk disease, and so is an appropriate agent for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and phenotypic verification of B cell CLL or SLL and measurable disease.
* Prior therapy: Patients must have been receiving single agent ibrutinib therapy at the time of disease progression. Patient may have received other therapy in combination with ibrutinib earlier in their treatment course.
* Women of childbearing potential (not postmenopausal for at least one year or not surgically incapable of bearing children) must agree not to become pregnant for the duration of the study.
* Adequate hematologic, hepatic and renal function

Exclusion Criteria:

* Known CNS lymphoma or leukemia
* History of Richter's or prolymphocytic transformation.
* Primary ibrutinib resistance
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenia purpura (ITP)
* History of major surgery within 4 weeks prior to first dose on this study.
* History of prior malignancy, with the exception of adequately treated non-melanoma skin cancer, malignancies treated with curative intent and with no evidence of active disease for more than 3 years, or adequately treated cervical carcinoma in situ without current evidence of disease.
* Active clinically significant cardiovascular disease or history of myocardial infarction within 6 months of first dose.
* Active hepatitis B or C infection.
* Known history of infection with human immunodeficiency virus (HIV).
* Unable to swallow capsules or disease significantly affecting gastrointestinal function.
* History of stroke or intracranial hemorrhage within 6 months of first dose.
* Requires anticoagulation with warfarin or other Vitamin K antagonists.
* Requires treatment with a strong cytochrome P(CYP)450 3A inhibitor.
* Pregnant or breast-feeding women
* Current infection requiring parenteral antibiotics.
* Active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification.
* Patients who require immediate cytoreduction due to high risk of tumor lysis syndrome (ie, absolute lymphocyte count greater than 100k/uL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose or biologically active dose. | 1 year or more
  Maximum tolerated dose or biologically active dose.

SECONDARY OUTCOMES:
Treatment-emergent adverse events | 2 years or more
  Treatment-emergent adverse events (description, timing, grade [CTCAE v4.03], severity, seriousness, and relatedness)
Overall response rate | 2 years or more
  Partial Response, Partial Response with Lymphocytosis, and Complete Response) based on international working group guidelines. Best overall response will be determined
Progression free survival rate at completion of combination therapy | 2 years or more
  Progression free survival rate at completion of combination therapy, duration of response, as determined by International Working Group in CLL (iwCLL) criteria.
Stable disease rate | 2 years or more
  Stable disease rate (also based on 2008 iwCLL guidelines), also at the time of primary endpoint response assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Choi, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States